CLINICAL TRIAL: NCT00482183
Title: Comparison of Bare Metal Stent With Pioglitazone Versus Sirolimus-Eluting Stent for Percutaneous Coronary Intervention in Patients With Type 2 Diabetes Mellitus.
Brief Title: Comparison Between Pioglitazone and SES With type2 DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Showa University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT-NAPN-16586; CCT-NAPN-16586
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Coronary Artery Disease; Type 2 Diabetes Mellitus
Keywords: Bare metal stent; Major adverse cardiac events; Pioglitazone; Restenosis; Sirolimus eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
Drug-eluting stents have been shown to decrease restenosis, but were associated with an increased rate of death, as compared with bare-metal stents. Recently, thiazolidinediones effectively reduced restenosis and the risk of repeat target vessel revascularization. We conducted a study to compare the performance of a drug-eluting stent with that of a bare-metal stent with pioglitazone in patients with type 2 diabetic mellitus.

DETAILED DESCRIPTION:
The study is a prospective cohort trial involving 38 type 2 diabetic patients referred for coronary stenting who were assigned to either the sirolimus-eluting stent group or the pioglitazone group. Quantitative coronary angiography will be performed at study entry and at six months follow-up to evaluate in-stent late luminal loss and the percentage of the luminal diameter and the rate of restenosis. We also analyze major adverse cardiac events at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who had received coronary stenting were eligible for the study.

Exclusion Criteria:

* spastic angina pectoris
* congestive heart failure
* hepatic dysfunction
* chronic renal disease
* recent stroke
* impaired glucose tolerance
* insulin dependent diabetes mellitus
* familial hypercholesterolemia
* thyroid dysfunction
* adrenal dysfunction
* an intolerance of aspirin, ticlopidine, heparin, pioglitazone, stainless steel, or contrast material.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary angiographic end point is in-stent luminal late loss, as determined by quantitative angiography. | Within 12minths after the procedure

SECONDARY OUTCOMES:
Secondary end points include the percentage of in-stent stenosis of luminal diameter, the rate of restenosis. | 6 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Youichi Kobayashi, Professor, Study Chair — Showa University

REFERENCES:
- [Derived] Nishio K, Shigemitsu M, Kodama Y, Konno N, Katagiri T, Kobayashi Y. Comparison of bare metal stent with pioglitazone versus sirolimus-eluting stent for percutaneous coronary intervention in patients with Type 2 diabetes mellitus. Cardiovasc Revasc Med. 2009 Jan-Mar;10(1):5-11. doi: 10.1016/j.carrev.2008.06.004. PMID 19159848